CLINICAL TRIAL: NCT03214471
Title: Evaluation of the Effect of a Lifestyle Intervention Compared to Usual Care on Weight Loss and Changes in Body Composition, Physical Activity Levels and Health-related Quality of Life in the First Year Following Bariatric Surgery
Brief Title: Evaluation of a Lifestyle Intervention After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16/0232
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Obesity
Keywords: bariatric surgery; healthy lifestyle
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The trial will be a two-arm, parallel group, single-blinded, single site RCT (embedded within an observational cohort study) conducted in London, United Kingdom (UK). A two-staged randomised consent design will be applied (See 8.2 Randomisation procedures). Recruitment will take place at the Bariatric Centre for Weight Management and Metabolic Surgery, University College London Hospitals (UCLH) and the Bariatric and Obesity Surgery Clinic at the Whittington Hospital. The trial will be carried out by the Centre for Obesity Research, Division of Medicine, University College London (UCL) at UCLH, which will be commenced in August 2017 with the expected total duration of 36 months. The total duration of each participation in the trial is approximately 12-16 months (12 months from the day of surgery). All participants will have to attend 4 research visits; baseline visit (approximately 6 weeks before surgery), then at approximately 3, 6, and 12-month post-surgery.
Who Masked: Outcomes Assessor
Masking Description: The investigator who will conduct the follow-up assessments at each visit will be blinded to participants' allocation and will not be involved in delivering any of the intervention. The statistician conducting the data analysis will be blind to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): usual care provided by the NHS for patients undergoing bariatric surgery.
- Intervention (Experimental): usual care + BARI-LIFESTYLE intervention
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Nutritional and behavioural tele-counselling , self-monitoring and a 12-week supervised tailored exercise programme. Participants will receive a regular tele-counselling throughout the 12-month. Each session will take approximately 15 minutes, underpinned by behavioural psychological techniques. After their 3-month post-surgery assessment visit, participants in the BARI-LIFESTYLE Intervention Study will be enrolled in a supervised exercise programme at health facility gyms for 12 weeks.
  Arms: Intervention

SUMMARY:
The aim of this trial is to evaluate the effect of a post-surgery 12-month lifestyle intervention compared to usual care upon post-surgery weight loss and changes that occur in body composition (relative amounts of body fat, muscle and bone), physical fitness and activity levels, diseases linked to obesity (e.g. diabetes, high blood pressure, high cholesterol level, sleep apnoea) and health-related quality of life (HRQoL) over a 12-month period.

DETAILED DESCRIPTION:
People with severe obesity who are scheduled to undergo either primary gastric bypass or primary sleeve gastrectomy will be recruited from the Bariatric Clinics at University College London Hospital (UCLH) and the Whittington Hospital and asked to participate in an observational cohort study. Eligible patients will be given a participant information sheet (PIS) for BARI-LIFESTYLE Observational Study and informed consent will be sought. Recruited patient will attend for 4 research visits, timed to coincide with their clinic visits, at approximately 6 weeks before surgery (Visit 1), 3 month post-surgery (Visit 2), 6 months post-surgery (Visit 3) and 12 months post-surgery (Visit 4). Each research visit will include assessment of body weight, body composition (using bioelectrical impedance analysis), physical fitness and activity levels, obesity-associated co-morbidities, HRQoL and usual care laboratory investigations. Dual energy X-ray absorptiometry (DXA) scanning will be undertaken at Visit 1 and Visit 4, which is not a usual assessment for the post-surgery standard care. All of the research assessments will be done as part of this observational cohort study.

Immediately after surgery has been undertaken, BARI-LIFESTYLE Observational Study participants will be randomised to continue to receive usual care, or usual care plus lifestyle intervention (nutritional and behavioural tele-counselling, self-monitoring and a 12-week supervised tailored exercise programme). However, to avoid contamination between the intervention group and the usual care group, only those randomly allocated to the lifestyle intervention group will be informed of this. They will be given a PIS (BARI-LIFESTYLE Intervention Study) and informed consent will be sought. If the participants decline to take part in the lifestyle programme, they will remain in the control group (observational cohort study).

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged between 18 to 65 years old.
2. Planned to undergo either primary gastric bypass surgery or primary sleeve gastrectomy surgery and fulfilling NICE eligibility criteria for bariatric surgery.
3. Medically safe to participate in exercise programme.
4. Able to read and write in English.
5. Willing and able to provide written informed consent.
6. Able to comply with study protocol.
7. Able to attend a supervised tailored exercise session at UCLH weekly for 12 weeks.
8. Willing and able to wear a Fitbit wrist-based activity tracker device and an Actigraph device.

Exclusion Criteria:

1. More than 200 kg of body weight (due to limitation of DXA Scanner).
2. Non-ambulatory.
3. Functional limitation.
4. Medical contraindication for exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
%WL | 52 weeks
  The primary objective of this trial is to compare the 1-year post-surgery percentage weight loss (%WL) in people receiving usual care and people receiving a post-operative lifestyle intervention programme.

SECONDARY OUTCOMES:
body fat | 52 weeks
  To compare post-surgery changes in body fat assessed using DXA scanning relative to pre-surgery at 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme.
bone mineral density | 52 weeks
  To compare post-surgery changes in bone mineral density assessed using DXA scanning relative to pre-surgery at 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme.
skeletal muscle mass | 52 weeks
  To compare post-surgery changes in skeletal muscle mass, relative to pre-surgery at 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme.
physical activity (PA) levels | 12, 26 and 52 weeks
  To compare post-surgery changes in physical activity (PA) levels (light, moderate, vigorous) at 3, 6, and 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme using Actigraph assessments.
150 minutes of activity | 12, 26 and 52 weeks
  To compare post-surgery changes in percentage achieving 150 minutes of moderate to vigorous PA (MVPA) in a week at 3, 6, and 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme using Actigraph assessments.
sedentary time | 12, 26 and 52 weeks
  To compare post-surgery changes in sedentary time at 3, 6, and 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme using Actigraph assessments.
6MWT | 12, 26 and 52 weeks
  To compare post-surgery changes in physical fitness assessed using 6-minute walk tests (6MWT) at 3, 6 and 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme.
STS | 12, 26 and 52 weeks
  To compare post-surgery changes in physical fitness assessed using sit-to-stand (STS) test at 3, 6 and 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme.
Handgrip test | 12, 26 and 52 weeks
  To compare post-surgery changes in handgrip test at 3, 6 and 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme.
36-Item Short-Form Health Survey Instrument (SF-36) | 12, 26 and 52 weeks
  To compare post-surgery changes in health-related quality of life.
Impact of Weight on Quality of Life-Lite (IWQOL-Lite) | 12, 26 and 52 weeks
  To compare post-surgery changes in health-related quality of life.
Beck Depression Inventory (BDI) | 12, 26 and 52 weeks
  To compare post-surgery changes in characteristics of attitude and symptoms of depression assessed using Beck Depression Inventory (BDI) at 3, 6 and 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme.
Medical history | 12, 26 and 52 weeks
  To compare post-surgery changes in obesity-associated comorbidities (type 2 diabetes, dyslipidaemia, hypertension, obstructive sleep apnoea) at 3, 6 and 12 months post-surgery in people receiving usual care and people receiving a post-operative lifestyle intervention programme.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Batterham, PhD FRCP, Principal Investigator — UCL
Locations (1):
- University College London Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
To be discussed

REFERENCES:
- [Background] Gloy VL, Briel M, Bhatt DL, Kashyap SR, Schauer PR, Mingrone G, Bucher HC, Nordmann AJ. Bariatric surgery versus non-surgical treatment for obesity: a systematic review and meta-analysis of randomised controlled trials. BMJ. 2013 Oct 22;347:f5934. doi: 10.1136/bmj.f5934. PMID 24149519
- [Background] Purnell JQ, Selzer F, Wahed AS, Pender J, Pories W, Pomp A, Dakin G, Mitchell J, Garcia L, Staten MA, McCloskey C, Cummings DE, Flum DR, Courcoulas A, Wolfe BM. Type 2 Diabetes Remission Rates After Laparoscopic Gastric Bypass and Gastric Banding: Results of the Longitudinal Assessment of Bariatric Surgery Study. Diabetes Care. 2016 Jul;39(7):1101-7. doi: 10.2337/dc15-2138. PMID 27289123
- [Background] National Clinical Guideline Centre (UK). Obesity: Identification, Assessment and Management of Overweight and Obesity in Children, Young People and Adults: Partial Update of CG43. London: National Institute for Health and Care Excellence (NICE); 2014 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK264165/ PMID 25535639
- [Background] Manning S, Pucci A, Carter NC, Elkalaawy M, Querci G, Magno S, Tamberi A, Finer N, Fiennes AG, Hashemi M, Jenkinson AD, Anselmino M, Santini F, Adamo M, Batterham RL. Early postoperative weight loss predicts maximal weight loss after sleeve gastrectomy and Roux-en-Y gastric bypass. Surg Endosc. 2015 Jun;29(6):1484-91. doi: 10.1007/s00464-014-3829-7. Epub 2014 Sep 20. PMID 25239175
- [Background] Tamboli RA, Hossain HA, Marks PA, Eckhauser AW, Rathmacher JA, Phillips SE, Buchowski MS, Chen KY, Abumrad NN. Body composition and energy metabolism following Roux-en-Y gastric bypass surgery. Obesity (Silver Spring). 2010 Sep;18(9):1718-24. doi: 10.1038/oby.2010.89. Epub 2010 Apr 22. PMID 20414197
- [Background] Giusti V, Theytaz F, Di Vetta V, Clarisse M, Suter M, Tappy L. Energy and macronutrient intake after gastric bypass for morbid obesity: a 3-y observational study focused on protein consumption. Am J Clin Nutr. 2016 Jan;103(1):18-24. doi: 10.3945/ajcn.115.111732. Epub 2015 Dec 16. PMID 26675775
- [Background] Janssen I, Fortier A, Hudson R, Ross R. Effects of an energy-restrictive diet with or without exercise on abdominal fat, intermuscular fat, and metabolic risk factors in obese women. Diabetes Care. 2002 Mar;25(3):431-8. doi: 10.2337/diacare.25.3.431. PMID 11874926
- [Background] Bond DS, Unick JL, Jakicic JM, Vithiananthan S, Pohl D, Roye GD, Ryder BA, Sax HC, Giovanni J, Wing RR. Objective assessment of time spent being sedentary in bariatric surgery candidates. Obes Surg. 2011 Jun;21(6):811-4. doi: 10.1007/s11695-010-0151-x. PMID 20393808
- [Background] Egberts K, Brown WA, Brennan L, O'Brien PE. Does exercise improve weight loss after bariatric surgery? A systematic review. Obes Surg. 2012 Feb;22(2):335-41. doi: 10.1007/s11695-011-0544-5. PMID 22038571
- [Background] Jassil FC, Manning S, Lewis N, Steinmo S, Kingett H, Lough F, Pucci AB, Cheung WH, Finer N, Walker J, Doyle J, Batterham RL. Feasibility and Impact of a Combined Supervised Exercise and Nutritional-Behavioral Intervention following Bariatric Surgery: A Pilot Study. J Obes. 2015;2015:693829. doi: 10.1155/2015/693829. Epub 2015 Jun 23. PMID 26199740
- [Background] Coen PM, Menshikova EV, Distefano G, Zheng D, Tanner CJ, Standley RA, Helbling NL, Dubis GS, Ritov VB, Xie H, Desimone ME, Smith SR, Stefanovic-Racic M, Toledo FG, Houmard JA, Goodpaster BH. Exercise and Weight Loss Improve Muscle Mitochondrial Respiration, Lipid Partitioning, and Insulin Sensitivity After Gastric Bypass Surgery. Diabetes. 2015 Nov;64(11):3737-50. doi: 10.2337/db15-0809. Epub 2015 Aug 20. PMID 26293505
- [Background] Sharman M, Hensher M, Wilkinson S, Williams D, Palmer A, Venn A, Ezzy D. What are the support experiences and needs of patients who have received bariatric surgery? Health Expect. 2017 Feb;20(1):35-46. doi: 10.1111/hex.12423. Epub 2015 Nov 2. PMID 28052539
- [Background] Pouwels S, Wit M, Teijink JA, Nienhuijs SW. Aspects of Exercise before or after Bariatric Surgery: A Systematic Review. Obes Facts. 2015;8(2):132-46. doi: 10.1159/000381201. PMID 25895670
- [Background] Bradley C. Designing medical and educational intervention studies. A review of some alternatives to conventional randomized controlled trials. Diabetes Care. 1993 Feb;16(2):509-18. doi: 10.2337/diacare.16.2.509. PMID 8432226
- [Background] Stott DJ, Langhorne P, Rodgers H. Informed consent. Two stage randomisation and consent would overcome many problems. BMJ. 1997 Jul 26;315(7102):253. No abstract available. PMID 9253294
- [Background] Zelen M. A new design for randomized clinical trials. N Engl J Med. 1979 May 31;300(22):1242-5. doi: 10.1056/NEJM197905313002203. PMID 431682
- [Background] Campbell R, Peters T, Grant C, Quilty B, Dieppe P. Adapting the randomized consent (Zelen) design for trials of behavioural interventions for chronic disease: feasibility study. J Health Serv Res Policy. 2005 Oct;10(4):220-5. doi: 10.1258/135581905774414150. PMID 16259688
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Beriault K, Carpentier AC, Gagnon C, Menard J, Baillargeon JP, Ardilouze JL, Langlois MF. Reproducibility of the 6-minute walk test in obese adults. Int J Sports Med. 2009 Oct;30(10):725-7. doi: 10.1055/s-0029-1231043. Epub 2009 Jul 7. PMID 19585400
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Pataky Z, Armand S, Muller-Pinget S, Golay A, Allet L. Effects of obesity on functional capacity. Obesity (Silver Spring). 2014 Jan;22(1):56-62. doi: 10.1002/oby.20514. Epub 2013 Aug 13. PMID 23794214
- [Background] O'Donovan G, Blazevich AJ, Boreham C, Cooper AR, Crank H, Ekelund U, Fox KR, Gately P, Giles-Corti B, Gill JM, Hamer M, McDermott I, Murphy M, Mutrie N, Reilly JJ, Saxton JM, Stamatakis E. The ABC of Physical Activity for Health: a consensus statement from the British Association of Sport and Exercise Sciences. J Sports Sci. 2010 Apr;28(6):573-91. doi: 10.1080/02640411003671212. PMID 20401789
- [Derived] Jassil FC, Carnemolla A, Kingett H, Doyle J, Kirk A, Lewis N, Montagut G, Marvasti P, Boniface D, Brown A, Chaiyasoot K, Zakeri R, Mok J, Devalia K, Parmar C, Batterham RL. Impact of nutritional-behavioral and supervised exercise intervention following bariatric surgery: The BARI-LIFESTYLE randomized controlled trial. Obesity (Silver Spring). 2023 Aug;31(8):2031-2042. doi: 10.1002/oby.23814. Epub 2023 Jul 6. PMID 37415246